CLINICAL TRIAL: NCT03033108
Title: A Phase 2a Multicenter, Randomized, Masked Study Evaluating the Pharmacodynamics of Emixustat Hydrochloride in Subjects With Macular Atrophy Secondary to Stargardt Disease
Brief Title: Pharmacodynamic Study of Emixustat Hydrochloride in Subjects With Macular Atrophy Secondary to Stargardt Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4429-204
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Stargardt Disease; Macular Atrophy
MeSH Terms: conditions — Stargardt Disease; Anetoderma | interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Emixustat Dose 1 (Experimental): lowest dose of once-daily oral emixustat
  Interventions: Drug: Emixustat
- Emixustat Dose 2 (Experimental): middle dose of once-daily oral emixustat
  Interventions: Drug: Emixustat
- Emixustat Dose 3 (Experimental): highest dose of once-daily oral emixustat
  Interventions: Drug: Emixustat

INTERVENTIONS:
Drug: Emixustat — Once daily, tablet for oral administration
  Other Names: emixustat hydrochloride

SUMMARY:
This is a pharmacodynamics study of emixustat hydrochloride in subjects with macular atrophy secondary to Stargardt disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, masked study to characterize the pharmacodynamics, safety and tolerability of emixustat in subjects with macular atrophy secondary to Stargardt disease.

ELIGIBILITY:
Inclusion Criteria, including, but not limited to:

* Clinical diagnosis of macular atrophy (MA) secondary to Stargardt disease (STGD) in one or both eyes
* At least 2 pathogenic mutations of the ABCA4 gene
* Early Treatment Diabetic Retinopathy Study BCVA of ≥ 20 letters (approximately ≥ 20/400 Snellen) in the study eye
* Adequate clarity of ocular media and adequate pupillary dilation to permit good quality imaging of MA in the study eye
* Able and willing to provide written informed consent before undergoing any study-related procedures
* Able to reliably administer oral medication by self or with available assistance

Exclusion Criteria, including, but not limited to:

* Macular atrophy associated with a condition other than STGD in either eye.
* Presence in either eye of an active ocular disease that in the opinion of the Investigator compromises or confounds visual function.
* History of any intraocular or ocular surface surgery in either eye within 3 months of screening.
* Current or previous participation in an interventional study to treat STGD using gene therapy or stem cell therapy at any time, or participation in an interventional study of a vitamin A derivative ≤3 months prior to screening.
* Pre-specified laboratory abnormalities at screening
* Presence of other medical or ophthalmic disease, physical examination finding, or clinical laboratory finding that in the opinion of the Investigator may contraindicate the use of an investigational drug and place the subject at risk
* Current or history of cancer (except for adequately treated basal cell or squamous cell carcinoma of the skin) within 1 year of screening
* History of myocardial infarction, stroke, unstable ischemic heart disease, uncontrolled cardiac arrhythmia, or hospitalization for congestive heart failure within 6 months of screening.
* Anticipated hospitalization for a medical/surgical procedure(s) that could result in interruption/premature cessation of study treatment or participation.
* Electrocardiogram with a clinically significant abnormal finding
* Female subjects who are pregnant or lactating
* Female subjects of childbearing potential or male subjects who are not surgically sterile who are not willing to practice a medically accepted method of birth control with their sexual partner from screening through 30 days after the final dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Acucela Medical Director, MD, Study Director — Kubota Vision Inc.
Locations (1):
- Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kubota R, Birch DG, Gregory JK, Koester JM. Randomised study evaluating the pharmacodynamics of emixustat hydrochloride in subjects with macular atrophy secondary to Stargardt disease. Br J Ophthalmol. 2022 Mar;106(3):403-408. doi: 10.1136/bjophthalmol-2020-317712. Epub 2020 Nov 19. PMID 33214244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 6 sites in the United States from January to September 2017
Period: Overall Study
Arm/Group | Emixustat Dose 1 | Emixustat Dose 2 | Emixustat Dose 3
Started | 7 | 9 | 7
Completed | 7 | 8 | 7
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emixustat Dose 1 | Emixustat Dose 2 | Emixustat Dose 3 | Total
Number analyzed (Participants) | 7 | 9 | 7 | 23
Age, Continuous [Mean (Full Range); unit: years] | 53.6 [27 to 77] | 54.3 [32 to 77] | 46.3 [18 to 70] | 51.6 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 3 | 8 | 4 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 9 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 5 | 7 | 6 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 7 | 23
Number of ABCA4 gene mutations [Count of Participants; unit: Participants]
  One mutation | 1 | 2 | 2 | 5
  Two mutations | 6 | 7 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Electrical Response of the Retina to a Flash of Light, as Measured by Electroretinogram
Description: Percent suppression compared to baseline of rod b-wave amplitude recovery after a photobleaching light.
Time Frame: Baseline and 1 month
Population: Subjects with evaluable ERGs at both Baseline and Month 1
Measure: Median (Full Range); unit: percent suppression
Arm/Group | Emixustat Dose 1 | Emixustat Dose 2 | Emixustat Dose 3
Number analyzed (Participants) | 6 | 7 | 6
percent suppression | -12.23 [-41.0 to 54.7] | 68.00 [1.0 to 91.5] | 96.69 [64.9 to 100.0]

2. Secondary Outcome: Percentage of Subjects With Adverse Events, by Severity and Seriousness
Description: Assessment of safety profile
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Emixustat Dose 1 | Emixustat Dose 2 | Emixustat Dose 3
Number analyzed (Participants) | 7 | 9 | 7
Participants
  Subjects with 1 or more adverse events | 6 | 8 | 6
  Subjects with 1 or more mild adverse events | 5 | 5 | 4
  Subjects with 1 or more moderate adverse events | 1 | 2 | 2
  Subjects with 1 or more severe adverse events | 0 | 1 | 1
  Subjects with 1 or more serious adverse events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Emixustat Dose 1 | Emixustat Dose 2 | Emixustat Dose 3
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 6/7 | 8/9 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Emixustat Dose 1 (N=7) | Emixustat Dose 2 (N=9) | Emixustat Dose 3 (N=7)
Delayed Dark Adaptation (Eye disorders) | 1 | 6 | 4
Erythropsia (Eye disorders) | 1 | 3 | 1
Vision blurred (Eye disorders) | 2 | 1 | 1
Photophobia (Eye disorders) | 1 | 2 | 0
Visual impairment (Eye disorders) | 1 | 1 | 1
Blindness day (Eye disorders) | 0 | 1 | 1
Chromatopsia (Eye disorders) | 0 | 0 | 2
Night blindness (Eye disorders) | 0 | 1 | 1
Xanthopsia (Eye disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2
Asthenopia (Eye disorders) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Eye Pain (Eye disorders) | 1 | 0 | 0
Eye Pruritis (Eye disorders) | 1 | 0 | 0
Lenticular opacities (Eye disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rhinorrheoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract infections (Infections and infestations) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Visual field defect (Nervous system disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Small sample size and inherent, significant intersubject and intrasubject variability observed in electroretinography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03033108/Prot_SAP_000.pdf